CLINICAL TRIAL: NCT04063085
Title: The Assessment of the Use of Anti-Adhesion Agents to Prevent Pelvic Postoperative Adhesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RDCT-TWPH
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-04

CONDITIONS: Tissue Adhesion; Gynecologic Surgery
Keywords: Hyaluronan; gel; adhesion agent
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PROTAHERE group (Experimental): The PROTAHERE group received intra-pelvic PROTAHERE Absorbable Adhesion Barrier during the scheduled pelvic surgery and be followed for 24 months.
  Interventions: Device: PROTAHERE Absorbable Adhesion Barrier
- Hyalobarrier group (Active Comparator): The Hyalobarrier group received intra-pelvic Hyalobarrier Gel during the scheduled pelvic surgery and be followed for 24 months.
  Interventions: Device: Hyalobarrier Gel
- No treatment group (Sham Comparator): The no treatment group did not receive any anti-adhesion agent during the scheduled pelvic surgery and be followed for 24 months.
  Interventions: Other: No treatment
- Seprafilm group (Active Comparator): The Seprafilm group received intra-pelvic Seprafilm Adhesion Barrier during the scheduled pelvic surgery and be followed for 24 months.
  Interventions: Device: Seprafilm Adhesion Barrier
- Interceed group (Active Comparator): The Interceed group received intra-pelvic Gynecare Interceed (TC7) Absorbale Adhesion Barrier during the scheduled pelvic surgery and be followed for 24 months.
  Interventions: Device: Gynecare Interceed (TC7) Absorbable Adhesion Barrier

INTERVENTIONS:
Device: PROTAHERE Absorbable Adhesion Barrier — 40 mg/ml (4%) cross-linked hyaluronan
  Arms: PROTAHERE group
Device: Hyalobarrier Gel — Laparotomy: 40 mg/ml (4%) cross-linked hyaluronan Endoscopy: 30 mg/ml (3%) cross-linked hyaluronan
  Arms: Hyalobarrier group
Other: No treatment — No anti-adhesion agent applied
  Arms: No treatment group
Device: Seprafilm Adhesion Barrier — a hyaluronate carboxymethylcellulose-based bioresorbable membrane
  Arms: Seprafilm group
Device: Gynecare Interceed (TC7) Absorbable Adhesion Barrier — an oxidized regenerated cellulose absorbable membrane
  Arms: Interceed group

SUMMARY:
The aim of this study is to assess the safety and effectiveness of PROTAHERE Absorbable Adhesion Barrier to prevent pelvic postoperative adhesions.

DETAILED DESCRIPTION:
The study is a random, evaluator-blinded, controlled, single center clinical trial. Recruiting patients who are premenopausal and scheduled for pelvic surgery including myomectomy, pelvic adhenolysis, endometriosis surgery, salpingostomy, dermoid cyst removal, ovarian cystectomy or any pelvic surgery other than total metrectomy. Patients recruited are randomly divided into five groups, PROTAHERE, Hyalobarrier, Seprafilm, Interceed or no treatment when the inclusion criteria are met and the inform consents are obtained. They are followed for 24 months including visits at 14 days, 3, 6, 12, 18, 24 months post-operation for the safety and effectiveness evaluation. The primary endpoints are the incidence of adhesions at 3-month as well as the incidence of any adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are premenopausal.
* Patients who are scheduled for pelvic surgery including myomectomy, pelvic adhenolysis, endometriosis surgery, salpingostomy, dermoid cyst removal, ovarian cystectomy or any pelvic surgery other than total metrectomy.
* Patients who are 20 years old or older.
* Patients who are able to understand the objectives, sign the informed consent form, and willing to comply with study procedures.

Exclusion Criteria:

* Patients who are 65 years old or older.
* Presence of uncontrolled diabetes, coagulative disorders, severe urinary system infection, or other severe diseases.
* Presence of malignant tumor or diagnosed with cancer.
* Any physical or psychological illness or symptom which is considered unsuitable to enroll by physicians.
* Patients who are unwilling to comply with study procedures.
* Patients who are known to have hypersensitivity to hyaluronic acid implants.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative adhesion at 3 months | 3 months post-operation
  Divide the number of patients with postoperative adhesion at 3 months in each group by the total number of patients enrolled.

SECONDARY OUTCOMES:
The incidence of adverse events in each group from the baseline and during the study period | 14 days, 3, 6, 12, 18, 24 months
  Divide the number of patients who suffered from adverse events by the number of patients enrolled in each group.
The incidence of each adverse event from the baseline and during the study | 14 days, 3, 6, 12, 18, 24 months
  Divide the number of each adverse event by the number of total adverse events.
The severity of adverse events | 14 days, 3, 6, 12, 18, 24 months
  The severity of adverse events are evaluated by blinded evaluators. The severity is classified into slight (no requirement for treatment), moderate (required for treatments, hospitalization or hospitalization prolongation) and serious (death, life-threatening, required for intensive care, required 7 days or longer time for recovery, permanent disability or congenital malformation)
The change of medication or treatment related to adverse event | 14 days, 3, 6, 12, 18, 24 months
  The change of time or dose of the medication or treatment in each group are evaluated by blinded evaluators.
The proportion of sites with adhesions at 3 months | 3 months post-operation
  Divide the number of sites with adhesions by the total number of sites observed.
The score of adhesion severity and extent at each sites at 3 months | 3 months post-operation
  Scoring method published by America Fertility Society:
  The score of filmy adhesions with less than 1/3 enclosure is 1. The score of filmy adhesions with 1/3-2/3 enclosure is 2. The score of filmy adhesions with more than 2/3 enclosure is 4. The score of dense adhesions with less than 1/3 enclosure is 4. The score of dense adhesions with 1/3-2/3 enclosure is 8. The score of dense adhesions with more than 2/3 enclosure is 16. Higher score indicates more severe and extent adhesions, and represents worse outcome.
The total score of America Fertility Society classifications of adhesions at all sites in each group at 3 months | 3 months post-operation
  Scoring method published by America Fertility Society:
  The score of filmy adhesions with less than 1/3 enclosure is 1. The score of filmy adhesions with 1/3-2/3 enclosure is 2. The score of filmy adhesions with more than 2/3 enclosure is 4. The score of dense adhesions with less than 1/3 enclosure is 4. The score of dense adhesions with 1/3-2/3 enclosure is 8. The score of dense adhesions with more than 2/3 enclosure is 16. The evaluated sites include anterior and posterior uterus, anterior and posterior cul-de-sac, left and right pelvic sidewall, left and right ovaries, left and right tubes, small bowel, large bowel, omentum, left and right abdominal wall as well as the incision, left and right broad ligament, left and right round ligament of uterus. Sum up all the adhesion scores at all sites in each group. The minimum total score is 0 and the maximum total score is 320. Higher score indicates more severe and extent adhesions, and represents worse outcome.
The incidence of postoperative adhesion from the baseline and during the study period | 14 days, 3, 6, 12, 18, 24 months
  Divide the number of patients with postoperative adhesion from the baseline and during the study in each group by the total number of patients enrolled.
The change of CA125 value in each group during the study period | 3, 6, 12, 18, 24 months
  CA125 value (U/ml) is considered as one of the indexes of pelvic inflammation.
The change of the results of SF-36 questionnaire in each group from the baseline and during the study period | 14 days, 3, 6, 12, 18, 24 months
  SF-36 questionnaires are filled out by patients to evaluate their health status during the study period. 8 categories of scales are evaluated including physical functioning, role limitations due to physical or emotional problems, energy/fatigue, emotional well beings, social functioning, pain and general health. For each category, the minimum average score is 0 and the maximum average score is 100. Higher score indicates better health status, which represents a better outcome.
The residual status of anti-adhesion agents at 3 months | 3 months post-operation
  The residual status of anti-adhesion agents at each site is evaluated by blinded evaluators. No residue is scored to be 0, and with residue is scored to be 1. Sum up the scores of all sites in each group.
Visual analog scale (VAS) score for pain change | 14 days, 3, 6, 12, 18, 24 months
  Patients enrolled who had endometriosis or intra-pelvic adhesions would subjectively evaluate their feeling of pain through a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain' during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan